CLINICAL TRIAL: NCT01349270
Title: Multicentre Randomized Open-label Trial to Compare Efficacy and Tolerance of Corticosteroids and IVIg in Patients With Chronic Inflammatory Demyelinating Polyneuropathy on a One Year Follow up
Brief Title: Randomized Open-label Trial to Compare Efficacy and Tolerance of Corticosteroids and IVIg
Acronym: PRNC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201084; 031213 (Other: AFSSAPS)
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Demyelinating Polyneuropathy
Keywords: chronic inflammatory demyelinating polyneuropathy; immunoglobulin; prednisone
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- immunoglobulin (Experimental): patient who received monthly 2g/kg cure of intravenous Immunoglobulin during 6 months
  Interventions: Drug: Immunoglobulin perfusion
- prednisone (Active Comparator): patient who received 0,8mg/kg/day of prednisone progressively tapered over 6 months
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Immunoglobulin perfusion — patient who received monthly 2g/kg intravenous cure of immunoglobulin
  Arms: immunoglobulin
Drug: Prednisone — patient who received 0,8mg/kg/day of prednisone progressively tapered over 6 months
  Arms: prednisone

SUMMARY:
Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) is a challenge because disease may generate important disability in patients including young adults. Randomized trials showed that corticosteroids, plasma exchanges and intravenous immunoglobulin (IVIg) can reduce impairment on a short term period but the treatment of a chronic disease doesn't agree with it. Corticosteroids and IVIg are the first line CIDP treatments. No study permits to demonstrate the superiority of one treatment to the other. Long term adverse effects of corticosteroids and IVIg cost are the respective limitation of their use. The investigators scheduled to recruit 40 CIDP patients in 23 French centres to receive either 0,8mg/kg/day of prednisone progressively tapered over 6 months or a monthly 2g/kg cure of IVIg during 6 months. Patients will be followed during 6 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 80, Weight ≤ 100 kg,

CIDP diagnosis:

* stable or deteriorated state (no spontaneous improvement),
* with the following features:
* motor or sensory and motor deficits, and reduced or abolished tendon reflexes,
* progressive or relapsing evolution,
* global symmetric disability in more than one limb,
* disease course installation over at least 2 months,
* cerebrospinal fluid with ≤10/µL white blood cells and > 0.5 g/L protein rate (non compulsory examination),
* electrophysiological or histological signs of demyelinization,
* INCAT disability score ≥ 2 in arms or ≥ 1 in legs

Exclusion Criteria:

* Severe electrophysiological axonal damage,
* Pure motor syndrome,
* Spontaneous improvement,
* Associated systemic disease that could be the cause of neuropathy,
* Severe cardiac insufficiency,
* Cardiac arrhythmia,
* Severe cardiopulmonary pathology,
* Inflammatory syndrome,
* Severe physical disease which can interfere with the trial,
* Patient in a strict salt-free diet,
* A clinically significant abnormal biological result,
* Positive serology in one of the following tests: HIV1, HIV2, A-B-C hepatitis, Hbs antigen, Lyme disease,
* IgA complete deficiency,
* History of anaphylactic reaction during previous IVIg infusion,
* Hypogammaglobulinemia (IgG < 3g/L),
* Creatinine clearance < 80 mL/min,
* Evolutive gastroduodenal ulcer, diabetes, serious infectious condition, evolutive virus disease (hepatite, herpes, varicella, zona), psychotic states not controlled by treatment, veinous or arterial thrombosis, non controlled high blood pressure, osteoporosis,
* Patient previously treated by corticosteroids, IVIg, plasma exchanges or any other immunosuppressive agent within 3 months before inclusion, except for azathioprine and mycophenolate mofetil which were tolerated in the case of the dose being unmodified within 3 months and kept unchanged during the trial,
* Experienced failure with a IVIG or prednisone prior treatment,
* Hypersensitivity to any components of the 2 treatments,
* Unsigned informed consent,
* Ongoing or planned pregnancy (mandatory pregnancy test at the screening visit), breastfeeding, effective contraception for over 3 months for women of childbearing age.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Main outcome | 3 months
  Rate of patients with a decreased INCAT score of at least 1 point after 3 months of treatment,
  * Responders: ≥ 1 point improvement in the INCAT score at 3 months in comparison to baseline,
  * Non responders: unchanged INCAT score at 3 months in comparison to baseline or patients for whom the primary endpoint can't be assessed because of the occurrence of an adverse event requiring treatment stop.

SECONDARY OUTCOMES:
Secondary outcome | 3 months
  Rate of cured patients i.e. INCAT score of 0 in legs and ≤ 1 in arms after 3, 6, 9 and 12 months,

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe CAMDESSANCHE, Dr, Principal Investigator — CHU de SAINT-ETIENNE
Locations (11):
- France (11):
  - CHU Clermont-Ferrand, Clermont-Ferrand, France
  - Chu Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Hôpital Neurologique de Lyon, Lyon
  - Chu Marseille, Marseille
  - Chu Nancy, Nancy
  - Chu Nantes, Nantes
  - CHU Nice, Nice
  - Chu Saint-Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Centre hospitalier de Valence, Valence

REFERENCES:
- [Derived] Bus SR, de Haan RJ, Vermeulen M, van Schaik IN, Eftimov F. Intravenous immunoglobulin for chronic inflammatory demyelinating polyradiculoneuropathy. Cochrane Database Syst Rev. 2024 Feb 14;2(2):CD001797. doi: 10.1002/14651858.CD001797.pub4. PMID 38353301